CLINICAL TRIAL: NCT00747591
Title: Correlation of Urine Concentration of S100B in Extremely Premature Infants With Gestational Age and Severity of Intraventricular Hemorrhage
Brief Title: Urine Concentration of S100B in Extremely Premature Infants
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Joanna Beachy Ph.D., M.D., University of Utah Neonatology
Other Study IDs: 10870
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Premature Infants
Keywords: urine; concentration; of S100B
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
S100B, a calcium-binding protein, is found predominantly in the central nervous system (CNS) and is increased in CSF and blood after CNS injury. There are two objectives to this study. Is urine S100B concentration correlated with the serum concentration of S100B in infants born at 29-36 weeks gestation. The presence and severity of intracranial pathology on S100B concentration will be investigated. Further analysis will demonstrate if birth weight, daily fluid intake, urine output, and urine creatinine influence this relationship.

DETAILED DESCRIPTION:
S100B is a low molecular weight calcium binding protein found predominantly in the central nervous system, specifically astroglial cells.[1] S100B plays a role in calcium-dependent information processing and intracellular is involved in the regulation of cytoskeleton and cell morphology.[1] S100B is secreted by astrocytes and exhibits dose dependent extracellular cytokine functions. In tissue culture at nanomolar concentration, S100B stimulates neuronal growth, development, and regeneration and protects against degeneration. At micromolar concentration, S100B is neurotoxic [2] and stimulates apoptosis potentially through interaction with RAGE receptor, by induction of NO synthase, and through the caspase cascade. Thus, markedly elevated concentration of S100B, released from damaged astrocytes, may propagate neuronal death. To support this hypothesis, over expression of S100B is present in wobble mice, an animal model for neuronal degeneration.[3] S100B is also increased in brains of patients with Alzheimer's disease [1] and in the amniotic fluid of fetuses [4] and brains of patients with Down's syndrome.[1]

S100B is released from damaged astroglial cells and may indirectly reflect neuronal damage.[5,6] S100B is elevated in cerebrospinal fluid (CSF) of adult patients within 48 hours after infarction and remains elevated for at least 7 days after the event.[6] S100B is also elevated in CSF for the first 3 days after traumatic brain injury [7] and subarachnoid hemorrhage.[8] S100B readily crosses a dysfunctional blood-brain barrier and serum concentration of S100B is significantly increased in adult patients after traumatic brain injury [9], stroke [10], or cardiac arrest.[5] Serum S100B rises for 2-4 days after brain trauma or infarct and its concentration correlates with size of damage as identified by CT scan. [9,10] For patients with traumatic brain injury, elevated concentration of S100B was noted on admission and significantly predicted development of increased intracranial pressure 4-5 days later. [9] After cardiac arrest, serum S100B concentration was statistically elevated by 30 minutes after initiation of CPR and continued to be significantly elevated in those patients who later exhibited brain damage by CT scan or neurological exam.[5] This significant elevation in serum S100B lasted for at least 7 days. In addition, serum S100B concentration correlated with morbidity [9] and neurological outcome. [10] While the t1/2 of S100B is ~2 hours in adults, persistent increased concentration of S100B in serum indicates continuous release from damaged cells.

S100B has been shown to be differentially distributed in different cortical regions of the brain during fetal development and increases in concentration during gestation, supporting its role in the development and maturation of the CNS.[11] It is postulated that early in development, S100B leads to glial cell proliferation while later it leads to extension of neurites, regulation of fiber sprouting, formation/maintenance of synapses, and maturation of glial cells.[1] Cord blood concentration of S100B has been shown to be inversely related to gestational age between 27 to 42 weeks gestation.[12] Thirty term infants (37-42 weeks) had cord blood S100B levels < 1 ug/L while 28 preterm infants (27-36 weeks) had cord blood levels between 0.5 and 2.7 ug/L. Higher serum concentration of S100B may be due to the lack of integrity of the blood-brain barrier in preterm infants in conjunction with an increased secretion of S100B from astroglial cells.

Due to its low molecular weight (10.5 kD) and high degree of solubility, S100B is excreted through the kidneys. It has been detected in the first void urine of infants between 26-42 weeks gestation with the most preterm infant exhibiting the highest concentration of S100B (3.17 ug/L). [13] Urine S100B concentration was at the detection limit of the assay (0.02 ug/L) for term infants. There was a significant negative correlation between S100B concentration in the urine and gestational age (r=-.79, p<0.001), but the data was not shown. Only 23 preterm infants (gestational age 26-36 weeks) were enrolled in the study and the average gestational age was not stated. Previous study from this laboratory demonstrated that urine S100B concentration did not significantly vary between 23-28 weeks gestation. {spr}

Infants with CNS injury have increased CSF, serum, and urine concentration of S100B. In asphyxiated term infants who later developed intracranial hemorrhage, S100B was shown to be elevated at 12 hours after birth when compared to asphyxiated term infants who did not develop intracranial pathology and to control term infants.[14] In another report, asphyxiated term infants, who at 3 months exhibited abnormal neurologic outcome or death, had markedly elevated S100B levels 12-24 hours after birth.[15] However, that study was limited by a small number of patients. Serum concentration of S100B was also significantly elevated (2.9 ug/L) in 8 term infants 3 days after initiating ECMO therapy. Daily cranial ultrasound evaluation identified intracranial hemorrhage in these infants by day 5-6. In other words, significant elevation of serum concentration of S100B occurred at least 2-3 days prior to ultrasound evidence of intracranial hemorrhage. Eight control infants, who also received ECMO therapy, had no ultrasonic evidence of intracranial hemorrhage and had no change in S100B above baseline (0.5 ug/L).[16]

The most common CNS trauma for preterm infants is intraventricular hemorrhage (IVH).[17] IVH originates in the microcirculation/capillary network of the germinal matrix. Altered cerebral blood flow secondary to poor cerebral autoregulation or systemic hypo- or hypertension, platelet and coagulation disturbances as seen in infection, and decreased capillary integrity and vascular support have been implicated in the pathogenesis of IVH. IVH is graded (1-4) by extent of hemorrhage seen by ultrasound. In grade I IVH, the blood is confined to the germinal matrix. In Grade II IVH, blood is present in the germinal matrix and a small of blood is present in the ventricles. Grade III IVH occurs when the ventricles are filled with blood and dilated. In Grade IV IVH, blood extends into the brain parenchyma due to venous congestion of the terminal veins that border the lateral ventricles which leads to white matter necrosis. Grades I and II IVH are not associated with an increase in developmental abnormalities, but do not insure normalcy. Grades III and IV IVH (severe IVH) are highly associated with developmental delay, specifically spastic hemiplegia affecting the lower extremities more than the upper extremities due to the proximity of the hemorrhage to the descending motor fibers, and may also affect intellect. IVH, both mild (grade 1-2) and severe (grade 3-4) are rarely seen in infants with gestational age > 28 weeks due to the developmental involution of vessels in the germinal matrix which is the source of this hemorrhage.[17]

S100B is elevated in CSF, serum and urine in preterm infants with IVH. S100B is elevated in CSF of preterm infants who had IVH and posthemorrhagic ventricular dilatation and subsequent neurologic disability at 12 months of age.[18] The timing of the ventricular tap was not specified or uniform and correlation between IVH and serum concentration of S100B was not determined. Serum concentration of S100B is increased in preterm infants (mean gestational age 35 weeks) with IVH (grade 1-4) when compared to preterm infants without IVH.[19] In this study, the highest serum level of S100B (5 ug/L) was noted in an infant who died. However, that study was complicated by a small number of patients (11 with IVH and 14 control infants), nonspecified range of gestational age, non-uniform blood sampling time (within the first 48 hours after birth), and grade 1 IVH seen in 50% of the infants.

Urine concentration of S100B in preterm infants (29-35 weeks) with IVH (grade 2-4) is elevated at birth and continues to increase over the subsequent 3 days when compared to control preterm infants.[20] The severity of IVH significantly correlated with the level of S100B in the urine. The highest level of S100B was seen in the five infants who died.

Previous studies from this laboratory have demonstrated that urine concentration of S100B was elevated in those infants with gestational age 23-28 weeks with severe (grade 3 or 4 IVH) when compared to control infants with no or grade 1 IVH on day 1. (SPR)

An important limitation of the above cited studies is insufficient numbers of neonates were studied to allow correlation of both gestational age and presence of severe IVH on either urine or serum S100B concentration. Most importantly, those studies involved preterm infants whose gestational age was > 27 weeks gestation. Severe IVH (grade 3-4) is rarely seen in infants who are > 28 weeks gestation. In addition, no report to date in adults, children, or infants has defined the relationship between urine and serum concentration of S100B. Furthermore, no report has clearly established baseline S100B concentration in infants with gestational age < 28 weeks. The specific aims of this study have been stated. If S100B concentration is significantly increased in infants with severe IVH, then S100B concentration may predict which infants are highly likely to develop severe IVH with ensuing significant morbidity and mortality and allow for early initiation of treatment to decrease extension of intracranial damage.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at <28 weeks gestation will be eligible for enrollment in this study.

Exclusion Criteria:

* Infants with fetal malformations, chromosomal anomalies, and clinically significant sepsis (retractable hypotension, neutropenia, and thrombocytopenia) will be excluded, other.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born at <28 weeks gestation will be eligible for enrollment in this study.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2002-11; Primary Completion 2005-02 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Beachy, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States